CLINICAL TRIAL: NCT04809909
Title: Effect of Peripheral Stimulation on Acupuncture Points for Pain Relief of Low Back Pain Patients - a Prospective, Double-blind Randomized Controlled Trial
Brief Title: Peripheral Stimulation of Acupuncture Points for Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chi-Wai Cheung, Head of Department and Clinical Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UW21-024
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: The randomization sequence will be generated by Microsoft Excel software. Blocked randomization will be done with an allocation ratio of 1:1 under block randomization (patients with lower back pain only or patient having low back pain with radicular pain). The assigned intervention group is stated in sequentially numbered, opaque, sealed envelopes, which will be opened by the attending therapist treating the patient. The investigator who is involved in sequence generation or allocation concealment will not be involved in enrolling participants or administering the intervention.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants, outcome assessors and data analysts will be kept blinded to the allocation status to avoid information bias. Patients who have no knowledge in acupuncture are told that the leads would be implanted at the acupuncture points that can be at or outside the painful sites. Only the pain physician administering the allocated intervention is unblinded, whereas he/she is not involved in data collection or analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peripheral stimulation of acupuncture points (PSAP) (Experimental): Two electrode leads will be implanted and connected to an external neurostimulator for electrical stimulation of acupuncture points.
  Interventions: Procedure: Peripheral stimulation of acupuncture points (PSAP)
- Peripheral nerve field stimulation (PNFS) (Active Comparator): Two electrode leads will be implanted and connected to an external neurostimulator for electrical stimulation of the painful area.
  Interventions: Procedure: Peripheral nerve field stimulation (PNFS)

INTERVENTIONS:
Procedure: Peripheral stimulation of acupuncture points (PSAP) — Electrode leads will be implanted at Bladder 25-bilateral (BL25), the acupoint commonly used for relief of chronic Low Back Pain in standardized acupuncture.
  Arms: Peripheral stimulation of acupuncture points (PSAP)
Procedure: Peripheral nerve field stimulation (PNFS) — Electrode leads will be implanted at the region of pain.
  Arms: Peripheral nerve field stimulation (PNFS)

SUMMARY:
For decades, chronic low back pain has been one of the major health complaints in Hong Kong. Without proper management, low back pain is associated with functional disability and decreased quality of life. However, currently, there is still no "gold standard" treatment for cure of the problem.

DETAILED DESCRIPTION:
Peripheral nerve field stimulation (PNFS) is a neuromodulation therapy which provides pain relief through electrical stimulation of the painful area at the lower back. Previous studies have shown that the use of PNFS is effective in reducing pain intensity and improving physical functioning.

Peripheral stimulation of acupuncture points (PSAP) is a novel therapeutic strategy which involves the combination of PNFS and acupuncture from traditional Chinese medicine. Through electrical stimulation of specific acupuncture points, synergistic effect and additional benefits such as relief of sciatica might be observed. As such, the intervention is of our interest in the study.

The study will involve 50 subjects. After signing the consent form, subjects will be randomly assigned to one of the two groups, either PSAP or PNFS.

For group PSAP, two electrode leads will be implanted and connected to an external neurostimulator for electrical stimulation of acupuncture points.

For group PNFS, two electrode leads will be implanted and connected to an external neurostimulator for electrical stimulation of the painful area.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has signed the Subject Informed Consent/Subject Information Sheet prior to randomization.
2. Patient is aged 18 or above at the time of informed consent.
3. Patient presents with chronic intractable non-specific, axial or radicular Low Back Pain.
4. Patient has had chronic pain for at least 6 months.
5. Patient presents with predominant back pain, with a back pain score of ≥ 5 on the 11-point Numerical Rating Scale (NRS).
6. For patients with radicular Low Back Pain, the severity of back pain is greater than or equal to that of leg pain.
7. In the opinion of the Principal Investigator, the patient's Low Back Pain is regarded as intractable, as defined by the failure of at least three different classes of Low Back Pain treatments (pharmaceutical and/or non-pharmaceutical).

Exclusion Criteria:

1. Patient has been or is currently being treated with spinal cord stimulation or an implantable intrathecal drug delivery system.
2. Patient has an implantable infusion pump or a cardiac pacemaker.
3. In the opinion of the Principal Investigator, the patient's painful area overlaps with the predetermined acupuncture point used in the study.
4. Patient has a life expectancy of less than one year.
5. Patient has an active psychiatric disorder that is likely to hinder assessment of pain-related outcomes and/or compliance with the study protocol.
6. Patient has a systemic infection or lupus erythematosus.
7. Patient has a history of coagulation disorder.
8. Patient has enrolled in or is planning to enrol in clinical trials that might confound the results of the study.
9. Patient is currently pregnant or planning to become pregnant in the following 12 months.
10. Patient has knowledge of acupuncture and knows the location of acupuncture sites for pain relief.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-11-05 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | at 2 weeks after procedure
  Patient rates the pain intensity on the eleven-point scale from 0 to 10, in which 0 represents an absense of pain while 10 indicates the worst imaginable pain。

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology, The University of Hong Kong, Hong Kong, China